CLINICAL TRIAL: NCT06862765
Title: Characterization and Outcomes of Patients Screened for Transcatheter Tricuspid Valve Replacement with LuX-Valve Via the Trans-jugular Vein Approach
Brief Title: Characterization and Outcomes of Patients Screened for Transcatheter Tricuspid Valve Replacement
Acronym: The TRI-RECRUI
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Jian Yang, Prof., Xijing Hospital
Other Study IDs: KY20192138
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: High-surgical Risk Patients with Severe Tricuspid Regurgitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TTVR Screening: In this study ,235 patients were screened successed for TTVR with LuX-Valve via the trans-jugular vein, and 105 patients were screend failed
  Interventions: Procedure: transcatheter tricuspid valve replacement

INTERVENTIONS:
Procedure: transcatheter tricuspid valve replacement — The LuX-valve was implanted under fluoroscopic and echocardiographic guidance via the transjugular vein approach. Once the delivery system was introduced, it was adjusted within the right heart chamber to be perpendicular to the tricuspid annulus. The anterior leaflet was grasped using two leaflet graspers, and the ventricular portion of the device component was gradually released. After deploying the atrial disc to ensure the elimination of TR, septal anchoring was performed, and the delivery system was subsequently withdrawn.

SUMMARY:
The TRI-RECRUIT Study was conducted of 340 consecutive patients for TTVR screening using LuX-Valve via the trans-jugular vein approach at seven cardiac centers. Patient-level clinical records, imaging dates and screening outcomes were retrospectively collected.

ELIGIBILITY:
Inclusion Criteria:

* (i) age > 18 years old; (ii) TR severity ≥ severe; (iii) New York Heart Association (NYHA) functional class ≥ Ⅱ; (iv) failed GDMT; (v) Euro-SCORE > 4.

Exclusion Criteria:

* (i) left ventricular ejection fraction < 40%; (ii) systolic pulmonary arterial pressure > 60 mmHg; (iii) prior TV surgery or left-sided valve surgery within the past 6 months; (iv) irreversible poor right ventricular function; (v) concomitant significant lesion needed for other major cardiac procedures or infective endocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 340 consecutive patients for TTVR screening using LuX-Valve Plus at seven cardiac centers.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
screening failure rate | baseline， postprocedural immediately，30 days postprocedurally，6 months postprocedurally，1 year postprocedurally

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital, Xiamen, Fujian
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Department of Cardiovascular Surgery, Xijing Hospital, Xi'an, Shaanxi
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No